CLINICAL TRIAL: NCT02150460
Title: A Comparison of One-site and Two-site Peribulbar Anaesthesia for Cataract Surgery at National Eye Centre, Kaduna. Nigeria
Brief Title: A Comparison of One-site and Two-site Peribulbar Anaesthesia for Cataract Surgery at Kaduna, Nigeria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Eye Centre, Kaduna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NECKAD/TRIALS/001/2012
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-05

CONDITIONS: Anaesthesia; Cataract
Keywords: ophthalmic surgery, peribulbar local anaesthesia
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-site peribulbar injection (Experimental): Injection of a mixture of lidocaine 2% + adrenaline 0.125mg/ml + hyaluronidase 15 International Units (IU)/ml into the inferior medial orbital compartment
  Interventions: Procedure: One-site peribulbar injection
- Two-site peribulbar injection (Active Comparator): Injection of a mixture of lidocaine 2% + adrenaline 0.125mg/ml + hyaluronidase 15IU/ml into the infero-temporal and supero-nasal orbital compartments
  Interventions: Procedure: Two- site peribulbar injection

INTERVENTIONS:
Procedure: One-site peribulbar injection — injection into the inferior medial orbital compartment
  Arms: One-site peribulbar injection
Procedure: Two- site peribulbar injection — Two injections into the infero-temporal and supero-nasal orbital compartments
  Arms: Two-site peribulbar injection

SUMMARY:
The aim of the study was to compare the efficacy and safety of single injection peribulbar anaesthesia against the classic double injection technique.

This was a double blind randomized controlled trial involving two groups of consenting, adult Nigerian subjects with operable age-related cataract. An anaesthetic nurse who allocated the subjects to the two groups administered all the injections. The same surgeon operated on all the subjects while the principal investigator and a research assistant measured the outcome variables. All others were blinded as to subject allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and above
* Diagnosed with uncomplicated senile cataract
* Visual acuity of <3/60

Exclusion Criteria:

* Impaired mental status
* Difficulty in speaking
* Known allergy to amide-type local anaesthetic agents and/ or hyaluronidase
* Previous surgery in the same eye
* Glaucoma
* Impaired ocular motility
* Eyelid abnormalities
* Patients with only one eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminatu A AbdulRahman, MBBS, FWACS, Principal Investigator — National Eye Centre, Kaduna; Mahmoud B Alhassan, MBBS, FWACS, Study Chair — National Eye Centre, Kaduna
Locations (1):
- National Eye Centre, Kaduna, Kaduna State, Nigeria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One-site Peribulbar Injection | Two-site Peribulbar Injection
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients aged 50 years and above with age related operable cataracts that presented for elective cataract surgery during the study period
Groups:
- Total: Total of all reporting groups
Arm/Group | One-site Peribulbar Injection | Two-site Peribulbar Injection | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.30 (7.4) | 62.60 (10.7) | 63.45 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 29 | 27 | 56
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 61.48 (13.0) | 57.38 (10.3) | 59.26 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Achieve Adequate Akinesia
Description: Time taken to achieve akinesia and anesthesia adequate for surgery. Ability to move the eye in each of four directions (up, down, right and left) was scored thus: 2- normal movement, 1- reduced movement and 0- flicker or no movement. Upper eyelid akinesia was scored as 2- normal opening, 1- reduced movement and 0- complete immobility. Maximum score of 10 and minimum of 0. Adequate akinesia was defined as a total score of <4 and was evaluated at 10 and 15 minutes.
Time Frame: 10 minutes and 15 minutes
Measure: Number; unit: participants
Groups:
- Group 1: One-site peribulbar injection
- Group 2: Two-site peribulbar injection
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
participants
  10 minutes | 41 | 41
  15 minutes | 9 | 9

2. Primary Outcome: Supplementary Injection(s)
Description: After 10 minutes if akinesia score was more than 3, supplementary injections were given and the effect assessed was 5 minutes later
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
participants | 9 | 9

3. Primary Outcome: Complications of Local Anaesthetic Injection
Description: Systemic complications: dyspnoea, bronchospasm, impaired consciousness, intravascular injection etc
  Local complications: eyelid oedema, corneal oedema, conjunctival chemosis, conjunctival haemorrhage, globe perforation, vitreous haemorrhage, orbital haemorrhage etc
Time Frame: 0,10 and 15 minutes
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
participants
  Deviation of the globe | 1 | 0
  Sunconjunctival haemorrhage | 0 | 1
  Chemosis | 0 | 14

4. Primary Outcome: Pain Score for Local Anaesthetic Injection
Description: Pain was scored using a 4 point scale: 1 - no pain, 2 - mild pain, 3 - moderate pain, 4 - severe pain
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
units on a scale | 1.64 (0.6) | 1.58 (0.6)

5. Secondary Outcome: Volume of Anaesthetic Drug (ml)
Description: Total volume of anaesthetic drug injected into the orbit to achieve anaesthesia and akinesia adequate for cataract surgery
Time Frame: 10 and 15 minutes
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
milliliters | 5.36 (0.78) | 5.40 (0.88)

6. Secondary Outcome: Total Number of Injections
Description: Total number of injections required to achieve an akinesia score of <4
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
injections | 1.18 (0.39) | 2.18 (0.39)

7. Secondary Outcome: Surgeon Satisfaction Score for Local Anaesthetic Block
Description: Surgeon subjectively scored satisfaction with the anaesthetic block on a 4 point scale: 1- poor (25%), 2 - fair (50%), 3 - good (75%), 4 - excellent (100%)
Time Frame: 20 minutes
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
units on a scale | 4 [1 to 4] | 4 [1 to 4]

8. Secondary Outcome: Acceptability of the Anaesthetic Block to the Subject
Description: Subjects were asked if they would agree to have the same anaesthetic procedure the next time they needed cataract surgery in the other eye
Time Frame: 25 minutes
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
participants | 50 | 50

9. Secondary Outcome: Duration of Cataract Surgery (Minutes)
Description: Time interval from conjunctival incision to application of eye pad
Time Frame: At the end of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
minutes | 8.78 (2.19) | 8.88 (2.40)

10. Primary Outcome: Pain Score for Cataract Surgery
Description: Pain was scored on a 4 point scale: 1 - no pain, 2 - mild pain, 3 - moderate pain, 4 - severe pain
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 50
units on a scale | 1.06 (0.2) | 1.06 (0.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 14/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=50) | Group 2 (N=50)
Chemosis (Eye disorders) | 0 (0) | 14 (14) — Swelling of the conjunctiva

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No